

# **Study Protocol**

Effects of low-intensity blood-flow restricted exercise compared to standard rehabilitation in patients with knee osteoarthritis - a randomized controlled trial

# **Trial registration**

ClinicalTrials.gov trial registration identifier:

Ethical Committee in Region Hovedstaden: H-19079135

Data Protection Agency: P-2019-814

## **Study Protocol Version and Date**

Version: 1.0

Date: 25.05.2022



# **Table of Contents**

| Background | 3 |
|----------------------------|---|
| Study Purpose | |
| Methods | |
| Inclusion criteria | |
| Exclusion criteria | |
| Outcome measures | |
| Statistical power analysis | 7 |
| Ethical considerations | |
| Practical conditions | 7 |
| References | 8 |



# **Background**

Osteoarthritis (OA) is the second most common disease in Denmark and it is estimated that over 1 million danish people suffer from OA in one or multiple joints<sup>1,2</sup>. A significant number of these people have to receive treatment to reduce pain and maintain the ability to work, and the socioeconomic costs in Denmark as a direct consequence of OA is estimated to be approximately 11 billion Danish kroner (1,5 million EUR) each year<sup>2</sup>.

Knee-OA is the most common OA-diagnosis and it is estimated that 60.000 Danish people with symptoms of knee-OA seek medical treatment each year<sup>3</sup>. The occurrence of knee-OA is related to overweight, inactivity, aging, earlier knee injuries and exposure to lifelong physical work<sup>4-6</sup>. The elderly population continuous to increase, and so does the numbers of inactive and overweight people and therefore the occurrence of knee-OA can be expected to increase in the coming decades.

Knee-OA patients often are offered a combination of patient education, weight loss counseling and physical exercise<sup>3,7</sup>. Physical exercise including conventional strength training, functional training (whole body exercises) and cardiovascular training all seem to have an beneficial effect on knee pain, functional function and quality of life in people with OA<sup>8-13</sup>. In Denmark, the GLA:D (Good Life with osteoArthritis in Denmark) concept is a nationwide exercise paradigm, which consists of eight weeks of designated and supervised multi-component training performed twice weekly<sup>14-16</sup>. The concept is a combination of education and supervised neuromuscular exercise (NEMEX) delivered by GLA:D-certified physiotherapists, with the purpose to improve lower limb muscle strength and increase muscular stability around the knee- and hip joints, respectively<sup>14-16</sup>. NEMEX has previously shown positive results on pain perception<sup>11,15-20</sup>, functional capacity<sup>11,15</sup> and quality of life<sup>15,16</sup>, however the effect of NEMEX (or GLA:D) on muscle strength and lower limb muscle mass has never been investigated to the best of our knowledge. Notably, deficits in maximal muscle strength is often a critical factor in people with knee-OA, and can reach of 20-40 % compared to healthy sex and age-matched individuals<sup>21-23</sup>. Furthermore, prior systematic reviews have indicated that reduced knee extensor muscle strength is an important risk factor for the incidence of KOA as well as for the severity of symptoms and the decline in functional performance<sup>5,24</sup>. As such, improving lower limb muscle strength, with a particular focus on knee extensor strength, may be a key factor in improving symptoms and function in KOA. People with OA, who are able to tolerate heavy strength training, typically experience a positive effect on maximal muscle strength and power<sup>25,26</sup>. Unfortunately however, a large proportion of OA patients are forced to refrain from this type of training due to excessive joint- and muscle pain during and following the training sessions<sup>27</sup>.



In recent years strength training combined with concurrent blood flow restriction, i.e. occlusion training, has gained increasing acceptance and usage in athletes<sup>28,29</sup> as well as different patient groups<sup>30-38</sup>. This type of training, often referred as BFR (Blood Flow Restricted) exercise, imposes low levels of mechanical stress on the involved muscles and joints because the exercises are performed with low training load (≤30% of max) concurrently with a reduced blood flow to the working muscles, which is achieved by means of a modified pneumatic blood pressure cuff. BFR training has been documented to result in significant improvements in muscle mass and muscle strength even with just a few weeks of intense daily training<sup>39-41</sup>. Moreover, especially in the clinical setting, BFR exercise has been reported to effectively activate muscular satellite cells (stem cells), which are involved in muscle regeneration and myofiber growth<sup>40,42</sup>. The marked improvements in muscle mass and strength with BFR training seem to be comparable to that achieved by conventionel heavy-resistance strength training<sup>31,34,37-39,43</sup>. Importantly, recent data indicate that BFR training can have an acute pain-reducing effect<sup>33,38</sup> and result in greater strength gains and more pronounced reductions in pain with daily activities compared to heavy strength training in knee patients who experiences pain during training<sup>30</sup>. Based on these observations BFR exercise may represent an attractive alternative training modality in patients with knee-OA.

# **Study Purpose**

To investigate whether an enhanced rehabilitating effect on muscle function and joint pain can be achieved by training with low-intensity BFR exercise compared to standard rehabilitation (education and exercise) in people with knee-OA.

#### **Methods**

Inclusion takes place via the Institute of Sports Medicine (ISMC), and the Department of Physical and Occupational Therapy at Bispebjerg Hospital, Copenhagen, Denmark. Assessment for inclusion is made after referral from general practitioner or after conversation with physician assessor at the ISMC. Recruitment will also include advertising through local newspapers, posters in public libraries etc., as well as invitations to attend lectures with information about the study.

Patients will be called in for an initial examination by the attending physicians. At the consultation a standard clinical assessment will be performed and the participant will be examined to ensure that they meet the explicit inclusion but have none of the exclusion criteria of the study. For participants that adhere to the inclusion criteria, an information document will be handed out and the participant will be invited to an in-depth interview regarding the study with a physician (FJ; clinical project leader and PI). Participants will be informed that they may bring a friend or family



member to the information interview. Standard radiographs will be obtained. An informed consent will be obtained if the patients meet all of the criteria. Randomization procedures will take place following baseline testing, and will be performed at Bispebjerg Hospital by a blinded (to group allocation) assessor. Subsequently, training intervention procedures will be initiated.

#### Inclusion criteria

- All participants must meet the American College of Rheumatology (ACR) criteria for OA<sup>44</sup>
- Visible OA on X-ray imaging (Kellgren & Lawrence grade 2-3)
- Pain and functional limited for a minimum of 3 months.
- Be able to voluntarily (i.e. unassisted) perform a 90 degrees flexion in the knee while standing
- Be able to perform loaded machine exercise (leg press and knee extension) planned for the BFR training.
- Be able to understand written and spoken Danish
- Be able to complete the intervention period without extensive time away.

#### Exclusion criteria

- Kellgren & Lawrence grade 1 and 4
- Bilateral OA-symptoms.
- Prior knee- or hip alloplasty.
- Glucocorticosteroid injection in the knee within the last 6 months.
- Inflammatory arthritis.
- Known neurotic disease such as multiple sclerosis or peripheral neuropathy.
- Prior myocardial infarct or stroke, or chest pain during physical activity.
- Other health related or medical conditions which makes it challenging to participate in the study.

Furthermore, it is an exclusion criterium in the following conditions where use of pneumatic occlusion would be considered contraindicated:

- Type I Diabetes
- Peripheral vascular disease
- Excessive varicose veins
- Prior history of deep venous thrombosis
- Venous insufficiens causing edema in the lower legs



• Systolic blood pressure over 160 mmHg or under 100 mmHg

All the included patients will be randomized into one of two intervention groups; education and neuromuscular exercise (GLA:D) or BFR training. Participants in the education and exercise group will be offered participation in the GLA:D programme<sup>16</sup>. The GLA:D training involve a circuit training program with four stations. Each station involves two to six exercises that the participants perform 10-15 repetitions over 2-3 sets, which depends on the participants pain- and functional level. The BFR group performs training with the knee-OA diagnosed leg. BFR training is performed with the BFR cuff placed at the top of the thigh on the leg being trained. The cuff will be inflated to 60-80 % of the total arterial occlusion pressure (AOP)<sup>45-49</sup>. The participant will then perform training of the knee extensors in a leg press exercise machine and a leg extension exercise machine with a load corresponding to 30 % of the maximal load (1RM = Repetition Maximum)<sup>46,47,49</sup>.

The intervention period will last 12 consecutive weeks with 2 weekly training sessions. The participants in the GLA:D group will attend a supervised group training with educated physiotherapy GLA:D instructors at several chosen physiotherapy clinics. Training in the BFR group will be conducted at Bispebjerg Hospital by trained supervisors who are experienced in BFR exercise intervention.

#### Outcome measures

Before the intervention period, all participants will be tested for a number of different outcome measures. The primary outcome variable is KOOS (Knee injury and Osteoarthritis Outcome Score) <sup>50,51</sup>. Secondary outcome variables at the functional level include maximal and habitual timed upand-go test (TUG)<sup>52</sup>, balance test of postural sway<sup>53</sup>, 30-s chair-stand test<sup>52</sup> and stair-climbing test<sup>52,54</sup>. Additional secondary outcome parameters related to mechanical muscle function and includes assessment of maximal knee extensor strength (KinCom, isokinetic dynamometer)<sup>55</sup>, explosive muscle strength (rate of force development, RFD) (KinCom, isokinetic dynamometer) <sup>55,56</sup>, maximal muscle power (Nottingham Power Rig) <sup>57</sup> and muscle mass (Ultrasonography and DXA-scan). Furthermore, muscle biopsies from the front thigh muscle (m. quadriceps) will be obtained in a sub-group (n=30) of patients for determination of selected myocellular parameters (fiber area, vascularization, muscular satellite cells, nuclei content)<sup>40,58,59</sup>. Testing will take place before the intervention period, after 8 weeks of training and at the end of the intervention (12 weeks) except for the muscle biopsies, which will take place before the intervention period and at the end (12 weeks).



Statistical power analysis

The estimated number of participants in the study are based on the primary outcome variable, KOOS, with the assumption that a chance of 10 KOOS points would be of clinical relevance as well as assuming a standard deviation (SD) of 15 points. With a statistical power of 80 %, a significance level of 0.05 and an expected change in KOOS of 10 point magnitude after 12 weeks of training, was calculated to require 37 participants. To account for drop outs, a total of 90 participants are planned to be included in the study.

### **Ethical considerations**

The study has been accepted by the Committees on Health Research Ethics in Region Hovedstaden (H-19079135). The study will be carried out in accordance with international, standardized research ethics considerations and has been approved by the Danish Data Protection Agency.

All outlined experimental methods have previously been used by the involved researchers at Bispebjerg Hospital (Institute of Sports Medicine and Geriatric Research Unit), Herlev Hospital (Geriatric Research Unit, Department of Internal Medicine) and University of Southern Denmark (Research Unit of Muscle Physiology and Biomechanics at the Department of Sport and Biomechanics), respectively. At no time previously have any serious incidents taken place in our facility that may contraindicate the usage of these methods involved in the present research study. Furthermore, there is no indications in the literature that patients with knee-OA cannot complete 12 weeks of BFR training<sup>25,26</sup>. Due to the low load and the controlled movements when using exercise machines in connection with BFR training, this form of exercise is generally well tolerated by OA patients, who also demonstrate a high training compliance to this training modality <sup>25,38</sup>. Finally, BFR training is not associated with risks of uncontrolled or pain-triggering movement patterns.

#### **Practical conditions**

The project will be completed at the Institute of Sports Medicine Copenhagen (ISMC) at Bispebjerg Hospital (BBH) where recruitment, testing, biopsy will be performed. Project activities (data analyses etc) will also be performed at the Institute of Sports Science and Clinical Biomechanics at the University of Southern Denmark, where all muscle biopsy laboratory analysis will be performed.



#### References

- 1. Jensen H, Davidsen M, Ekholm O, Christensen A. Danskernes Sundhed Den Nationale Sundhedsprofil 2021. *Sundhedsstyrelsen*. 2022;
- 2. Johnsen N, Kock M, Davidsen M, Juel K. De samfundsmæssige omkostninger ved artrose. *Statens Institut for Folkesundhed*. 2014;
- 3. Sundhedsstyrelsen. Knæartrose Nationale kliniske retningslinjer og faglige visitationsretningslinjer. 2012;
- 4. Ashkavand Z, Malekinejad H, Vishwanath BS. The pathophysiology of osteoarthritis. *Journal of Pharmacy Research*. 2013/01/01/ 2013;7(1):132-138. doi:https://doi.org/10.1016/j.jopr.2013.01.008
- 5. Øiestad BE, Juhl CB, Eitzen I, Thorlund JB. Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis.

  Osteoarthritis and cartilage. 2015;23(2):171-177. doi:10.1016/j.joca.2014.10.008
- 6. Silverwood V, Blagojevic-Bucknall M, Jinks C, Jordan JL, Protheroe J, Jordan KP. Current evidence on risk factors for knee osteoarthritis in older adults: a systematic review and meta-analysis. *Osteoarthritis and cartilage*. Apr 2015;23(4):507-15. doi:10.1016/j.joca.2014.11.019
- 7. McAlindon TE, Bannuru RR, Sullivan MC, et al. OARSI guidelines for the non-surgical management of knee osteoarthritis. *Osteoarthritis and cartilage*. Mar 2014;22(3):363-88. doi:10.1016/j.joca.2014.01.003
- 8. Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. *BMC musculoskeletal disorders*. Jun 17 2010;11:126. doi:10.1186/1471-2474-11-126
- 9. Dantas LO, Salvini TF, McAlindon TE. Knee osteoarthritis: key treatments and implications for physical therapy. *Braz J Phys Ther*. Mar-Apr 2021;25(2):135-146. doi:10.1016/j.bjpt.2020.08.004
- 10. Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: A Cochrane Systematic Review. *Br J Sports Med.* Jan 9 2015;1:1554-7. doi:10.1002/14651858.CD004376.pub3
- 11. Holm PM, Schrøder HM, Wernbom M, Skou ST. Low-dose strength training in addition to neuromuscular exercise and education in patients with knee osteoarthritis in secondary care a randomized controlled trial. *Osteoarthritis and cartilage*. Jun 2020;28(6):744-754. doi:10.1016/j.joca.2020.02.839



- 12. Skou ST, Rasmussen S, Laursen MB, et al. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. *Osteoarthr Cartil*. Sep 2015;23(9):1465-75. doi:10.1016/j.joca.2015.04.021
- 13. Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. *The Journal of rheumatology*. Jul 2014;41(7):1385-94. doi:10.3899/jrheum.130642
- 14. Roos EM, Grønne DT, Skou ST, et al. Immediate outcomes following the GLA:D® program in Denmark, Canada and Australia. A longitudinal analysis including 28,370 patients with symptomatic knee or hip osteoarthritis. *Osteoarthr Cartil*. Apr 2021;29(4):502-506. doi:10.1016/j.joca.2020.12.024
- 15. Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. *Danish medical journal*. Dec 2012;59(12):A4554.
- 16. Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D™): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. *BMC musculoskeletal disorders*. Feb 7 2017;18(1):72. doi:10.1186/s12891-017-1439-y
- 17. Bandak E, Christensen R, Overgaard A, et al. Exercise and education versus saline injections for knee osteoarthritis: a randomised controlled equivalence trial. *Ann Rheum Dis.* Nov 29 2021;doi:10.1136/annrheumdis-2021-221129
- 18. Davis AM, Kennedy D, Wong R, et al. Cross-cultural adaptation and implementation of Good Life with osteoarthritis in Denmark (GLA:D™): group education and exercise for hip and knee osteoarthritis is feasible in Canada. *Osteoarthritis and cartilage*. Feb 2018;26(2):211-219. doi:10.1016/j.joca.2017.11.005
- 19. Holm PM, Petersen KK, Wernbom M, Schrøder HM, Arendt-Nielsen L, Skou ST. Strength training in addition to neuromuscular exercise and education in individuals with knee osteoarthritis-the effects on pain and sensitization. *Eur J Pain*. Oct 2021;25(9):1898-1911. doi:10.1002/ejp.1796
- 20. Skou ST, Bricca A, Roos EM. The impact of physical activity level on the short- and long-term pain relief from supervised exercise therapy and education: a study of 12,796 Danish patients with knee osteoarthritis. *Osteoarthritis and cartilage*. Nov 2018;26(11):1474-1478. doi:10.1016/j.joca.2018.07.010



- 21. Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. *Rheumatic diseases clinics of North America*. Aug 2008;34(3):731-54. doi:10.1016/j.rdc.2008.05.005
- 22. Rodriguez-Lopez C, Beckwée D, Luyten FP, Van Assche D, Van Roie E. Reduced knee extensor torque production at low to moderate velocities in postmenopausal women with knee osteoarthritis. *Scand J Med Sci Sports*. Nov 2021;31(11):2144-2155. doi:10.1111/sms.14035
- 23. Skoffer B, Dalgas U, Mechlenburg I, Soballe K, Maribo T. Functional performance is associated with both knee extensor and flexor muscle strength in patients scheduled for total knee arthroplasty: A cross-sectional study. *Journal of rehabilitation medicine*. May 2015;47(5):454-9. doi:10.2340/16501977-1940
- 24. Culvenor AG, Ruhdorfer A, Juhl C, Eckstein F, Øiestad BE. Knee Extensor Strength and Risk of Structural, Symptomatic, and Functional Decline in Knee Osteoarthritis: A Systematic Review and Meta-Analysis. *Arthritis care & research*. May 2017;69(5):649-658. doi:10.1002/acr.23005
- 25. Bryk FF, Dos Reis AC, Fingerhut D, et al. Exercises with partial vascular occlusion in patients with knee osteoarthritis: a randomized clinical trial. *Knee surgery, sports traumatology, arthroscopy.* May 2016;24(5):1580-6. doi:10.1007/s00167-016-4064-7
- 26. Ferraz RB, Gualano B, Rodrigues R, et al. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. *Medicine and science in sports and exercise*. May 2018;50(5):897-905. doi:10.1249/mss.000000000001530
- 27. Jan MH, Lin JJ, Liau JJ, Lin YF, Lin DH. Investigation of clinical effects of high- and low-resistance training for patients with knee osteoarthritis: a randomized controlled trial. *Physical therapy*. Apr 2008;88(4):427-36. doi:10.2522/ptj.20060300
- 28. Manimmanakorn A, Hamlin MJ, Ross JJ, Taylor R, Manimmanakorn N. Effects of low-load resistance training combined with blood flow restriction or hypoxia on muscle function and performance in netball athletes. *Journal of science and medicine in sport*. Jul 2013;16(4):337-42. doi:10.1016/j.jsams.2012.08.009
- 29. Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Blood flow restricted exercise for athletes: A review of available evidence. *Journal of science and medicine in sport*. May 2016;19(5):360-7. doi:10.1016/j.jsams.2015.04.014
- 30. Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. *Br J Sports Med.* Dec 2017;51(23):1688-1694. doi:10.1136/bjsports-2016-096329



- 31. Grønfeldt BM, Lindberg Nielsen J, Mieritz RM, Lund H, Aagaard P. Effect of bloodflow restricted vs heavy-load strength training on muscle strength: Systematic review and meta-analysis. *Scand J Med Sci Sports*. May 2020;30(5):837-848. doi:10.1111/sms.13632
- 32. Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. *Br J Sports Med.* Jul 2017;51(13):1003-1011. doi:10.1136/bjsports-2016-097071
- 33. Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. *Journal of applied physiology (Bethesda, Md : 1985)*. Apr 1 2020;128(4):914-924. doi:10.1152/japplphysiol.00768.2019
- 34. Lixandrão ME, Ugrinowitsch C, Berton R, et al. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. *Sports medicine* (Auckland, NZ). Feb 2018;48(2):361-378. doi:10.1007/s40279-017-0795-y
- 35. Takada S, Okita K, Suga T, et al. Low-intensity exercise can increase muscle mass and strength proportionally to enhanced metabolic stress under ischemic conditions. *Journal of applied physiology (Bethesda, Md : 1985)*. Jul 2012;113(2):199-205. doi:10.1152/japplphysiol.00149.2012
- 36. Yasuda T, Fukumura K, Fukuda T, et al. Muscle size and arterial stiffness after blood flow-restricted low-intensity resistance training in older adults. *Scand J Med Sci Sports*. Oct 2014;24(5):799-806. doi:10.1111/sms.12087
- 37. Dos Santos LP, Santo R, Ramis TR, Portes JKS, Chakr R, Xavier RM. The effects of resistance training with blood flow restriction on muscle strength, muscle hypertrophy and functionality in patients with osteoarthritis and rheumatoid arthritis: A systematic review with meta-analysis. *PloS one*. 2021;16(11):e0259574. doi:10.1371/journal.pone.0259574
- 38. Rodrigues R, Ferraz RB, Kurimori CO, et al. Low-Load Resistance Training With Blood-Flow Restriction in Relation to Muscle Function, Mass, and Functionality in Women With Rheumatoid Arthritis. *Arthritis care & research*. Jun 2020;72(6):787-797. doi:10.1002/acr.23911
- 39. Centner C, Wiegel P, Gollhofer A, König D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. *Sports medicine (Auckland, NZ)*. Jan 2019;49(1):95-108. doi:10.1007/s40279-018-0994-1



- 40. Nielsen JL, Aagaard P, Bech RD, et al. Proliferation of myogenic stem cells in human skeletal muscle in response to low-load resistance training with blood flow restriction. *The Journal of physiology*. Sep 1 2012;590(17):4351-61. doi:10.1113/jphysiol.2012.237008
- 41. Ramos-Campo DJ, Scott BR, Alcaraz PE, Rubio-Arias JA. The efficacy of resistance training in hypoxia to enhance strength and muscle growth: A systematic review and meta-analysis. *European journal of sport science*. Feb 2018;18(1):92-103. doi:10.1080/17461391.2017.1388850
- 42. Jakobsgaard JE, Christiansen M, Sieljacks P, et al. Impact of blood flow-restricted bodyweight exercise on skeletal muscle adaptations. *Clinical physiology and functional imaging*. Feb 15 2018;doi:10.1111/cpf.12509
- 43. Kubo K, Komuro T, Ishiguro N, et al. Effects of low-load resistance training with vascular occlusion on the mechanical properties of muscle and tendon. *J Appl Biomech*. May 2006;22(2):112-9.
- 44. Altman R, Asch E, Bloch D, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. *Arthritis and rheumatism*. Aug 1986;29(8):1039-49. doi:10.1002/art.1780290816
- 45. Clarkson MJ, May AK, Warmington SA. Is there rationale for the cuff pressures prescribed for blood flow restriction exercise? A systematic review. *Scand J Med Sci Sports*. Aug 2020;30(8):1318-1336. doi:10.1111/sms.13676
- 46. Næss T. Determining the optimal blood flow restriction protocol for maximising muscle hypertrophy and strength, pressure and cuff width: A mini-review. *J Hum Sport Exerc*. 01/01 2020;16doi:10.14198/jhse.2021.164.02
- 47. Patterson SD, Hughes L, Head P, Warmington S, Brandner C. Blood flow restriction training: a novel approach to augment clinical rehabilitation: how to do it. *Br J Sports Med*. Dec 2017;51(23):1648-1649. doi:10.1136/bjsports-2017-097738
- 48. Patterson SD, Hughes L, Warmington S, et al. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Review. *Front Physiol*. 2019-May-15 2019;10(533)doi:10.3389/fphys.2019.00533
- 49. Vanwye WR, Weatherholt AM, Mikesky AE. Blood Flow Restriction Training: Implementation into Clinical Practice. *Int J Exerc Sci.* 2017;10(5):649-654.
- 50. Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee



Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). *Arthritis care & research*. Nov 2011;63 Suppl 11:S208-28. doi:10.1002/acr.20632

- 51. Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS) development of a self-administered outcome measure. *The Journal of orthopaedic and sports physical therapy*. Aug 1998;28(2):88-96. doi:10.2519/jospt.1998.28.2.88
- 52. Dobson F, Hinman RS, Roos EM, et al. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. *Osteoarthritis and cartilage*. Aug 2013;21(8):1042-52. doi:10.1016/j.joca.2013.05.002
- 53. Sturnieks DL, Arnold R, Lord SR. Validity and reliability of the Swaymeter device for measuring postural sway. *BMC Geriatr*. 2011;11:63-63. doi:10.1186/1471-2318-11-63
- Suetta C, Magnusson SP, Rosted A, et al. Resistance Training in the Early Postoperative Phase Reduces Hospitalization and Leads to Muscle Hypertrophy in Elderly Hip Surgery Patients—A Controlled, Randomized Study. *Journal of the American Geriatrics Society*. 2004/12/01 2004;52(12):2016-2022. doi:10.1111/j.1532-5415.2004.52557.x
- Suetta C, Aagaard P, Rosted A, et al. Training-induced changes in muscle CSA, muscle strength, EMG, and rate of force development in elderly subjects after long-term unilateral disuse. *Journal of applied physiology (Bethesda, Md : 1985)*. Nov 2004;97(5):1954-61. doi:10.1152/japplphysiol.01307.2003
- Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. *Journal of applied physiology (Bethesda, Md : 1985)*. Oct 2002;93(4):1318-26.

  doi:10.1152/japplphysiol.00283.2002
- 57. Caserotti P, Aagaard P, Larsen JB, Puggaard L. Explosive heavy-resistance training in old and very old adults: changes in rapid muscle force, strength and power. *Scand J Med Sci Sports*. Dec 2008;18(6):773-82. doi:10.1111/j.1600-0838.2007.00732.x
- 58. Mertz KH, Reitelseder S, Jensen M, et al. Influence of between-limb asymmetry in muscle mass, strength, and power on functional capacity in healthy older adults. *Scand J Med Sci Sports*. Dec 2019;29(12):1901-1908. doi:10.1111/sms.13524



59. Nielsen JL, Frandsen U, Jensen KY, et al. Skeletal Muscle Microvascular Changes in Response to Short-Term Blood Flow Restricted Training-Exercise-Induced Adaptations and Signs of Perivascular Stress. *Frontiers in physiology*. 2020;11:556. doi:10.3389/fphys.2020.00556